CLINICAL TRIAL: NCT00971282
Title: Adjunctive Usage of a Moisturizing Lotion (Cetaphil® Moisturizing Lotion) to Limit the Skin Irritation Linked to the Set-up of a Treatment by Topical Retinoid (Differin® Gel 0,1%) in Healthy Subjects of Chinese Origins
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: RD.03.SPR.29076
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Results first posted 2012-05-15 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2012-04

CONDITIONS: Healthy Skin
MeSH Terms: interventions — cetyl alcohol, propylene glycol, sodium lauryl sulfate non-lipid cleansing lotion

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- intra-individual comparison (Experimental)
  Interventions: Drug: adapalen 0.1%; Other: Cetaphil®

INTERVENTIONS:
Drug: adapalen 0.1% — Intra-individual (split-face) comparison: Differin® 0.1% (whole face) will be applied once daily for 4 weeks.
  Visits will be conducted weekly for a maximum of 5 visits.
Other: Cetaphil® — Intra-individual (split-face) comparison: Cetaphil® (only one side of the face) will be applied once daily for 4 weeks.
  Visits will be conducted weekly for a maximum of 5 visits.

SUMMARY:
This is a single-center study, randomized, Investigator/Evaluator-blinded bilateral (split-face) comparison.

The objective: To assess the benefit of the concomitant use of a Moisturizing Lotion in reducing the skin irritation induced by a adapalen gel treatment in Chinese Subjects.

DETAILED DESCRIPTION:
The interest & relevance of the concomitant use of a non-comedogenic moisturizer in order to decrease retinoid irritation has already been demonstrated in Caucasian patients. Such interest of associating a moisturizer when Differin® gel is prescribed has not been demonstrated in Asian populations.

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects of Chinese origins
* aged 21 years or older
* with healthy skin;

Exclusion Criteria:

* skin pigmentation which interferes with the reading of skin reactions
* with sunburn, eczema, atopic dermatitis, perioral dermatitis, or rosacea on the area to be treated
* with a washout period for the following topical treatment(s) Corticosteroids, oher anti-inflammatory drugs, retinoids
* with a washout period for the following systemic treatment(s): Medications that may increase photosensitivity, corticosteroids, anti-inflammatories, retinoids

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr LEOW, Principal Investigator — National Skin Center
Locations (1):
- national Skin Center, Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Groups:
- Intra-individual Comparison: Differin applied once daily (evening) on the whole face Cetaphil applied once daily (morning) on 1 side of the face
Period: Overall Study
Arm/Group | Intra-individual Comparison
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intra-individual Comparison
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 10
Region of Enrollment [Number; unit: participants]
  Singapore | 30

OUTCOME MEASURES:

1. Primary Outcome: Erythema Rating Scale
Description: score from 0 (none) to 3 (severe)
Time Frame: at 4 weeks
Population: safety population (APT)
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Cetaphil + Differin: Differin applied once daily (evening) Cetaphil applied once daily (morning)
- Differin Alone: Differin applied once daily (evening)
Arm/Group | Cetaphil + Differin | Differin Alone
Number analyzed (Participants) | 30 | 30
units on a scale | 0.6 (0.7) | 0.7 (0.7)

2. Primary Outcome: Scaling
Description: score from 0 (none) to 3 (severe)
Time Frame: at 4 weeks
Population: safety population (APT)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cetaphil + Differin | Differin Alone
Number analyzed (Participants) | 30 | 30
units on a scale | 0.3 (0.6) | 0.6 (0.8)

3. Primary Outcome: Dryness
Description: score from 0 (none) to 3 (severe)
Time Frame: at 4 weeks
Population: safety population (APT)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cetaphil + Differin | Differin Alone
Number analyzed (Participants) | 30 | 30
units on a scale | 0.3 (0.5) | 0.4 (0.6)

4. Primary Outcome: Stinging/Burning
Description: score from 0 (none) to 3 (severe)
Time Frame: at 4 weeks
Population: safety population (APT)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cetaphil + Differin | Differin Alone
Number analyzed (Participants) | 30 | 30
units on a scale | 0.5 (0.6) | 0.6 (0.6)

5. Primary Outcome: Pruritus
Description: score from 0 (none) to 3 (severe)
Time Frame: at 4 weeks
Population: safety population (APT)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cetaphil + Differin | Differin Alone
Number analyzed (Participants) | 30 | 30
units on a scale | 0.5 (0.6) | 0.6 (0.7)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: All medical clinical events occurred after subject's consent signature and during the study, whether observed by the Evaluator/Injector or reported by the Subject and whether or not thought to be treatment-related were considered adverse events and collected.
Groups:
- Cetaphil + Differin; Differin Alone: intra-individual comparison
Arm/Group | Cetaphil + Differin | Differin Alone
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 10/30 | 10/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetaphil + Differin (N=30) | Differin Alone (N=30)
dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (3)
excoriation (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
scab (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
skin exfoliation (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any intent of the investigator to publish or disclose in any way the information requires the sponsor's prior written approval. The investigator shall provide their draft of such publication to sponsor for review and approval at least 2 months prior to the date of the intended publication. Sponsor shall have the absolute right to determine whether information may be published by the investigator.